CLINICAL TRIAL: NCT05544994
Title: The Effect of Aerobic Exercise Training in Patients With Type III Spinal Muscular Atrophy"
Brief Title: The Effect of Aerobic Exercise Training in Patients With Type III Spinal Muscular Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, sezanmergen, Msc -Physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aerobic Training
Record Dates: First submitted 2022-08-19; First posted 2022-09-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neuromuscular Diseases; Spinal Muscular Atrophy Type 3
Keywords: Spinal Muscular Atrophy Type 3; Aerobic Training; SMN protein level; Physiotherapy
MeSH Terms: conditions — Neuromuscular Diseases; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Training Group (Experimental): Aerobic training will be performed 3 days a week for 12 weeks at 60% -%75 of their maximum hearth rate with 30 minutes total duration consisting of 5 min warm up and 5 min cool down period in treatment group.
  Home exercise program will be given. This home program will include stretching, breathing, normal joint movement for 3 to 5 days a week
  Interventions: Other: Aerobic Exercise Training; Other: Home exercise program
- Control Group (Active Comparator): Home exercise program will be given. This home program will include stretching, breathing, normal joint movement, for 3 or 5 days a week.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Aerobic Exercise Training — Aerobic training will be performed 3 days a week for 12 weeks at 60%-%75 of their maximum hearth rate with 30 minutes total duration consisting of 5 min warm up and 5 min cool down period in treatment group.
  Arms: Aerobic Exercise Training Group
Other: Home exercise program — Home exercise program will be given. This home program will include stretching, breathing, normal joint movement, for 3 to 5 days a week.

SUMMARY:
In the last 10-15 years, a better understanding of the pathophysiology and molecular genetics of SMA has led to the emergence of previously unavailable pharmacological and genetic treatments.One of these new treatments, Nusinersen, targets SMN2, which is a slightly different copy of SMN1, and increases SMN protein levels.

Preclinical studies have provided evidence that neuroprotection is strongly formed, with exercise significantly increasing motor neuron survival independent of SMN expression.

In a limited number of clinical studies prior to Nusinersen treatment, it was reported that aerobic exercise training improved maximum oxygen uptake (VO2 max) without causing muscle damage, but still caused fatigue.

The aim of this study is to determine the effect of aerobic exercise training on motor and respiratory functions, exercise capacity, fatigue and quality of life in SMA Type III patients who can walk and receive Nusinersen therapy. Twenty cases aged 10-50 years with genetically confirmed SMA diagnosis will be included in this study. The cases to be included in the study will be randomized into 2 groups as the training and control groups.

In addition to the routine physiotherapy program, medium-intensity Aerobic Exercise Training will be given to the study group for 12 weeks. Before and 12 weeks after the training, the cases will be evaluated with the Six Minute Walking Test, Submaximal Exercise Test, SMN protein level, function and strength assessments, (FVC) value, fatigue and quality of life scales.

In clinical trials, the supporting evidence for aerobic interventions in SMA is limited.

Additional studies on aerobic intervention parameters (frequency, intensity and duration) are needed.The results of this study will determine the feasibility of aerobic exercise training and provide important guidance for the clinical management of SMA patients.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a neuromuscular disorder characterized by degeneration of alpha motor neurons in the spinal cord, leading to progressive muscle atrophy and weakness. Mutation or deletion of the survival motor neuron1 (SMN1) gene causes insufficient production of the SMN protein, which ensures motor neuron survival and maintenance in the spinal cord.

In the last 10-15 years, a better understanding of the pathophysiology and molecular genetics of SMA has led to the emergence of previously unavailable pharmacological and genetic treatments. One of these new treatments, Nusinersen targets SMN2, which is a slightly different copy of SMN1, increases SMN protein levels. Preclinical studies have provided evidence that exercise significantly increases motor neuron survival independent of SMN expression, and that neuroprotection is strongly formed. In a limited number of clinical studies prior to Nuinersen therapy, it was reported that aerobic exercise training improved maximum oxygen uptake (VO2 max) without causing muscle damage, but still caused fatigue and had no significant beneficial effect on physical functioning. This study aims to determine the effect of aerobic exercise training on motor and respiratory functions, exercise capacity, fatigue and quality of life in SMA Type III patients who can walk and receive Nusinersen treatment. Twenty patients between the ages of 10 and 50 with genetically confirmed SMA diagnosis will be included in this study. The patients will be randomly divided into 2 groups as the training and control groups. In addition to the routine physiotherapy program, the study group will be given a moderate-intensity Aerobic Exercise Training for 12 weeks. Before and after 12 weeks of training, subjects will be evaluated with the Six-Minute Walk Test, ,Submaximal Exercise Test, SMN protein level and function and strength assessments, (FVC) value, fatigue and quality of life scales.

In clinical trials, the supporting evidence for aerobic interventions in SMA is limited. It has been reported that SMA patients cannot tolerate excessive exercise intensity and that recovery may be prevented due to excessive fatigue. Additional studies on aerobic intervention parameters (frequency, intensity and duration) are needed. The results of this study will determine the feasibility of aerobic exercise training and will have an impact on clinical practice by providing important guidance to the clinical management of SMA patients.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed of SMA Type 3 confirmed by genetic analysis,
* Between the ages of 10-50,
* Being able to walk 25 m without assistive device

Exclusion criteria:

* Using research drugs for SMA treatment other than Nusinersen treatment,
* Having a serious systemic disease that may prevent exercise,
* Have had a lower extremity injury and/or surgery in the last 6 months,
* To be applying a regular aerobic training program in the last 6 months

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | Baseline and 12 weeks
  Change from baseline functional capacity test at 12 weeks. Functional capacity will be assessed by the 6 minute walking test.The 6MWT, an objective evaluation of functional capacity, measures the maximum distance a person can walk in six minutes over a 25-meter linear course.

SECONDARY OUTCOMES:
Submaximal Exercise Test | Baseline and 12 weeks
  Change from baseline Submaximal Exercise Capacity Test at 12 weeks. It will be evaluated by Incremental Submaximal Exercise Test. The tests will be performed by using an cycle ergometer.
Pulmonary Function | Baseline and 12 weeks
  Change from baseline Forced Vital Capacity (FVC) in respiratory function test at 12 weeks. Pulmonary Function will be assessed by measuring forced expiratory vital capacity (FVC) as percent predicted for age and height.
Motor Function | Baseline and 12 weeks
  Change from baseline Hammersmith Functional Motor Scale, Expanded (HFMSE) at 12 weeks . The HFMSE is a 33-item scale designed for SMA type 2 and 3 patients.Items are scored on a 0-2 scale with a full score of 2 being normal without assistance, a partial score of 1 requiring a modified method but no assistance, and a zero score being unable to achieve the task without assistance.
Motor Performance | Baseline and 12 weeks
  Change from baseline 10 Meter Walk/Run Test at 12 weeks . This test measures the time it takes a subject to walk or run 10 meters as fast as possible without compromising the subject's safety.
Balance and Mobility | Baseline and 12 weeks
  Change from baseline Timed Up and Go Test (TUG) Test at 12 weeks The TUG test, which is a method to assess balance and mobility, measures the time it takes an individual to stand up from a chair, walk 3 meters, turn around, and sit down in the same chair.Ten seconds or less indicate normal mobility.
Muscle strength | Baseline and 12 weeks
  Change from baseline Manual Muscle Testing (MMT) at 12 weeks Manual muscle testing (MMT) augmented by hand held dynamometry (HHD) provides a comprehensive evaluation of muscle strength.
Quality of Life in patients with neuromuscular disease | Baseline and at 12 weeks
  Change from baseline quality of life scale at 12 weeks The Pediatric quality of life™ 3.0 Neuromuscular Module (PedsQL™ 3.0 NMM) was designed to assess health-related quality of life (HRQoL) among aged 2-18 years with NMD.The scale consists of 25 items under 3 categories. .Items are scored on a Likert-type scale from 0 (never poses a problem) to 4 (always poses a problem). Scoring is between 0-100 .Higher scores from the Module indicate better health-related quality of life.For patients 18 years and older, The Short Form (SF-36), a widely used health-related quality of life measure. The Short Form (SF-36) Health Survey is a 36-item, patient-reported survey of patient health.
Fatigue | Baseline and 12 weeks
  Change from baseline Fatigue Scale at 12 weeks.
  The PedsQL Multidimensional Fatigue Scale comprises parallel child self-report and parent proxy-reportformats. A 5-point response scale is utilized across child and a dolescent self-report for ages 8-18 and paren proxy-report .
  Items are reverse scored and linearly transformed to a 0-100 scale.Higher PedsQL Multidimen-sional Fatigue Scale scores indicate better HRQOL.
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in adult patients with a variety of disorders .A self-report scale of nine items about fatigue,The higher the score, the more severe the fatigue is and the more it affects the person's activities.
Functional Lower Extremity Strength, | Baseline and 12 weeks
  Change from baseline Five Times Sit to Stand Test at 12 weeks.
  The five Times Sit to Stand Test( 5XSS) scoring is based on the amount of time a patient is able to transfer from a seated to a standing position and back to sitting five times.
  The lower the time to complete the test the better the outcome of the test. The Minimal Detectable Change(MDC) time for the test is within 3.6 to 4.2 second and Minimal clinically important difference (MCID) is 2.3 seconds.
Evaluation of SMN protein levels in blood biochemistry | Baseline and 12 weeks
  Change from baseline SMN protein levels at 12 weeks. The response of patients' SMN protein levels to exercise will be evaluated before and after 12 weeks of training.

CONTACTS AND LOCATIONS:
Overall Officials: Sezan Mergen KILIÇ, MSc PT, Principal Investigator — Istanbul University, Istanbul Faculty of Medicine,Department of Neurological Sciences; Fatma Karantay Mutluay,, Professor, Study Director — Medipol University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Fatma Yeşim Parman, Professor, Study Director — Istanbul University, Istanbul Faculty of Medicine,Department of Neurological Sciences
Locations (1):
- Istanbul Faculty of Medicine, Department of Neurological Sciences, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No